CLINICAL TRIAL: NCT00003108
Title: A Phase I Study of Bryostatin and Cisplatin in Patients With Advanced Cancer
Brief Title: Cisplatin Plus Bryostatin 1 in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lombardi Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: GUMC-97166; CDR0000065849 (Registry Identifier: PDQ (Physician Data Query)); NCI-T97-0056
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2004-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — bryostatin 1; Cisplatin

INTERVENTIONS:
Drug: bryostatin 1
Drug: cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of cisplatin plus bryostatin 1 in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the dose limiting toxicity and maximum tolerated dose of combination bryostatin 1 and cisplatin chemotherapy in patients with advanced, incurable solid tumors.

OUTLINE: This is a dose-escalation study. The first 4 cohorts of patients receive an escalating dose of cisplatin with a fixed dose of bryostatin 1, followed by 5 cohorts receiving an escalating dose of bryostatin 1 and a fixed dose of cisplatin. In the first course, cisplatin is given as a 2 hour infusion followed by a 24 hour continuous infusion of bryostatin 1. In all subsequent courses bryostatin 1 is given first and cisplatin afterwards. Treatment continues every 21 days in patients with stable or responding disease. Dose escalation proceeds until the maximum tolerated dose (MTD) of the combination chemotherapy is determined. The MTD is defined as the dose preceding that at which 2 or more patients experience dose limiting toxicity. After the MTD is determined, an additional 10 patients are treated at this dose level. Patients are followed at 1 month.

PROJECTED ACCRUAL: Approximately 24-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, incurable solid tumor that is unresectable or has distant metastasis for which a more effective therapy does not exist No active CNS metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 8 weeks Hematopoietic: WBC at least 3000/mm3 Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL Transaminases no greater than 2.5 times normal PT and PTT no greater than 1.25 times upper limit of normal Renal: Creatinine no greater than 1.4 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: No myocardial infarction within past 6 months No congestive heart failure or serious arrhythmias requiring treatment Other: No greater than grade 2 neuropathy (including hearing loss) No frequent vomiting or severe anorexia No recent loss of greater than 10% of body weight Not pregnant or nursing Fertile patients must use effective birth control during and for at least 6 months after study No serious concurrent medical illness that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered from toxic effects No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (at least 6 weeks since prior mitomycin or nitrosoureas) and recovered No other concurrent chemotherapy Endocrine therapy: Concurrent hormonal therapy allowed if patient has progressive disease while receiving hormonal therapy for at least three months Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiation therapy Surgery: At least 21 days since prior major surgery Other: Any drugs that affect hepatic or renal function must be given as a stable dose and should not be initiated after patient enters study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-10; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L. Marshall, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (1):
- Lombardi Cancer Center, Washington D.C., District of Columbia, United States